CLINICAL TRIAL: NCT04326790
Title: The GReek Study in the Effects of Colchicine in Covid-19 cOmplications Prevention
Acronym: GRECCO-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment as a result of the rapid flattening of the curve of COVID-19 cases in Greece
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Spyridon Deftereos, Professor of Cardiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 906295542
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Corona Virus Disease 19 (Covid 19)
MeSH Terms: conditions — COVID-19 | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Patient-level randomization scheme
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Colchicine, on top of standard treatment
  Interventions: Drug: Colchicine; Drug: Standard treatment
- Control (Active Comparator): Standard treatment, including all medications recommedned by the National Public Health Organization
  Interventions: Drug: Standard treatment

INTERVENTIONS:
Drug: Colchicine — Low-dose colchicine treatment, 0.5 mg bid
  Arms: Intervention
Drug: Standard treatment — Standard treatment

SUMMARY:
Based on data regarding the effect of colchicine on the inflammasome NLP3 and microtubule formation and associations thereof with the pathogenetic cycle of SARS-COV-2, the question arises whether colchicine, administered in a relatively low dose, could potentially have an effect the patients' clinical course by limiting the myocardial necrosis and pneumonia development in the context of COVID-19. If present, this effect would be attributed to its potential to inhibit inflammasome and (less probably) to the process of SARS-CoV-2 endocytosis in myocardial and endothelial respiratory cells.

ELIGIBILITY:
Inclusion Criteria:

Patients >18 years old with laboratory confirmed SARS-CoV-2 infection (RT PCR) AND body temperature >37.5 degrees centigrade AND at least two of: i. sustained coughing, ii. sustained throat pain, iii. anosmia and/or ageusia, iv. fatigue/tiredness, v. PaO2<95 mmHg.

Exclusion Criteria:

* pregnancy, lactation;
* known hypersensitivity to colchicine
* known hepatic failure
* eGFR<20 ml/min
* clinical estimation that the patient will require mechanical respiratory support in less than 24 hours
* any clinical estimation of the attending physician under which the patient shall be excluded
* QTc > 450 msec (colchicine is not known to significantly prolong QTc, but may interact with other medications which prolong QTc).
* participation in another clinical trial
* under colchicine treatment for other indications
* patient who is not likely to comply to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Clinical deterioration in the semiquantitative ordinal scale suggested by the WHO R&D committee | 3 weeks
  Time to clinical deterioration (2 levels in the WHO R&D Blueprint scale)
Maximal concentration of cardiac troponin | 10 days
  Maximal concentration of high-sensitivity cardiac troponin

CONTACTS AND LOCATIONS:
Locations (1):
- National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014
- [Derived] Deftereos SG, Giannopoulos G, Vrachatis DA, Siasos GD, Giotaki SG, Gargalianos P, Metallidis S, Sianos G, Baltagiannis S, Panagopoulos P, Dolianitis K, Randou E, Syrigos K, Kotanidou A, Koulouris NG, Milionis H, Sipsas N, Gogos C, Tsoukalas G, Olympios CD, Tsagalou E, Migdalis I, Gerakari S, Angelidis C, Alexopoulos D, Davlouros P, Hahalis G, Kanonidis I, Katritsis D, Kolettis T, Manolis AS, Michalis L, Naka KK, Pyrgakis VN, Toutouzas KP, Triposkiadis F, Tsioufis K, Vavouranakis E, Martinez-Dolz L, Reimers B, Stefanini GG, Cleman M, Goudevenos J, Tsiodras S, Tousoulis D, Iliodromitis E, Mehran R, Dangas G, Stefanadis C; GRECCO-19 investigators. Effect of Colchicine vs Standard Care on Cardiac and Inflammatory Biomarkers and Clinical Outcomes in Patients Hospitalized With Coronavirus Disease 2019: The GRECCO-19 Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e2013136. doi: 10.1001/jamanetworkopen.2020.13136. PMID 32579195
- [Derived] Deftereos SG, Siasos G, Giannopoulos G, Vrachatis DA, Angelidis C, Giotaki SG, Gargalianos P, Giamarellou H, Gogos C, Daikos G, Lazanas M, Lagiou P, Saroglou G, Sipsas N, Tsiodras S, Chatzigeorgiou D, Moussas N, Kotanidou A, Koulouris N, Oikonomou E, Kaoukis A, Kossyvakis C, Raisakis K, Fountoulaki K, Comis M, Tsiachris D, Sarri E, Theodorakis A, Martinez-Dolz L, Sanz-Sanchez J, Reimers B, Stefanini GG, Cleman M, Filippou D, Olympios CD, Pyrgakis VN, Goudevenos J, Hahalis G, Kolettis TM, Iliodromitis E, Tousoulis D, Stefanadis C. The Greek study in the effects of colchicine in COvid-19 complications prevention (GRECCO-19 study): Rationale and study design. Hellenic J Cardiol. 2020 Jan-Feb;61(1):42-45. doi: 10.1016/j.hjc.2020.03.002. Epub 2020 Apr 3. PMID 32251729